CLINICAL TRIAL: NCT02301117
Title: A Phase 1, Open-Label Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of TAS-102 in Patients With Advanced Solid Tumors and Varying Degrees of Renal Impairment
Brief Title: A Phase I Study of TAS-102 in Patients With Advanced Solid Tumors With Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Taiho Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TO-TAS-102-107
Record Dates: First submitted 2014-11-13; First posted 2014-11-25 (Estimated); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Advanced Solid Tumors
Keywords: Renal; Kidney Diseases; Urologic Diseases; Renal Insufficiency; Renal Impairment; Pharmacokinetics; Advance Solid Tumor; Creatinine Clearance; Kidney Neoplasms; Renal Tumor; Kidney; Urology; Pharmacologic Action
MeSH Terms: conditions — Kidney Diseases; Urologic Diseases; Renal Insufficiency; Kidney Neoplasms; Carcinoma, Renal Cell | interventions — trifluridine tipiracil drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Mild Renal Impairment (Experimental): 35 mg/m2/dose of TAS-102 orally, twice daily on days 1-5 and days 8-12 of each 28 day cycle. Number of cycles: approximately 4 or until discontinuation criteria is met.
  Interventions: Drug: TAS-102
- Moderate Renal Impairment (Experimental): 35 mg/m2/dose of TAS-102 orally, twice daily on days 1-5 and days 8-12 of each 28 day cycle. Number of cycles: approximately 4 or until discontinuation criteria is met.
  Interventions: Drug: TAS-102
- Severe Renal Impairment (Experimental): 35 mg/m2/dose of TAS-102 orally, twice daily on days 1-5 and days 8-12 of each 28 day cycle. Number of cycles: approximately 4 or until discontinuation criteria is met.
  The dose level of severe cohort will be determined based on the Interim Assessment of mild and moderate cohorts
  Interventions: Drug: TAS-102
- Normal Renal Function (Experimental): 35 mg/m2/dose of TAS-102 orally, twice daily on days 1-5 and days 8-12 of each 28 day cycle. Number of cycles: approximately 4 or until discontinuation criteria is met.
  Interventions: Drug: TAS-102

INTERVENTIONS:
Drug: TAS-102

SUMMARY:
Study to evaluate the safety, tolerability, and pharmacokinetics of TAS-102 in patients with advanced solid tumors and varying degrees of renal impairment.

DETAILED DESCRIPTION:
This is a Phase 1, open-label study to evaluate the safety, tolerability, and pharmacokinetics of TAS-102 in patients with advanced solid tumors with varying degrees of renal impairment. The study is conducted in 2 parts: the Pharmacokinetic Part (Cycle 1) and the Extension Part (Cycles 2 and beyond). Patients may continue to receive treatment with TAS-102 during the study extension part only after completion of the Pharmacokinetic Part.

ELIGIBILITY:
Inclusion

1. Has provided written informed consent
2. Has advanced solid tumors (excluding breast cancer)
3. Has normal renal function, mild, moderate, or severe renal impairment and is not on dialysis
4. ECOG performance status of ≤2
5. Is able to take medications orally
6. Has adequate organ function
7. Women of childbearing potential must have a negative pregnancy test and must agree to adequate birth control if conception is possible. Males must agree to adequate birth control.

Exclusion

1. Certain serious illnesses or medical condition(s)
2. Has had certain other recent treatment e.g. major surgery, anticancer therapy, extended field radiation, received investigational agent, within the specified time frames prior to study drug administration
3. Has received TAS-102
4. Has unresolved toxicity of greater than or equal to CTCAE Grade 2 attributed to any prior therapies
5. Is a pregnant or lactating female

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2019-06-19 (Actual); Study Completion 2019-06-19 (Actual)

PRIMARY OUTCOMES:
PK parameters of FTD, FTY, and TPI in plasma after a single dose of TAS-102 | Blood samples will be collected in Cycle 1 Day 1 and Day 12 at pre-dose, 0.5, 1, 2, 4, 6, 8, 10, and 12 hours post AM dose of TAS-102
  FTD, FTY and TPI: pharmacokinetic parameters Cmax, Tmax, AUC0-last, AUC0-inf, and T1/2. FTD, FTY, and TPI: Ae% and CLr. FTD and TPI: CL/F, Vd/F of TAS-102
Safety monitoring including adverse events, vital signs, and laboratory assessments | Through 30 days following last administration of study medication or until initiation of new anticancer treatment

CONTACTS AND LOCATIONS:
Locations (13):
- United States (9):
  - Phoenix Clinical Site, Phoenix, Arizona
  - Duarte Clinical Site, Duarte, California
  - Santa Monica Clinical Site, Santa Monica, California
  - Gainesville Clinical Site, Gainesville, Florida
  - Baltimore Clinical Site, Baltimore, Maryland
  - Boston Clinical Site, Boston, Massachusetts
  - Cleveland Clinical Site, Cleveland, Ohio
  - Pittsburgh Clinical Site, Pittsburgh, Pennsylvania
  - Dallas Clinical Site, Dallas, Texas
- Czechia (2):
  - Brno Clinical Site, Brno
  - Praha Clinical Site, Prague
- Serbia (2):
  - Belgrade Clinical Site, Belgrade
  - Sremska Kamenica Clinical Site, Kamenitz

REFERENCES:
- [Derived] Saif MW, Becerra CR, Fakih MG, Sun W, Popovic L, Krishnamurthi S, George TJ, Rudek MA, Shepard DR, Skopek J, Sramek V, Zaric B, Yamamiya I, Benhadji KA, Hamada K, He Y, Rosen L. A phase I, open-label study evaluating the safety and pharmacokinetics of trifluridine/tipiracil in patients with advanced solid tumors and varying degrees of renal impairment. Cancer Chemother Pharmacol. 2021 Sep;88(3):485-497. doi: 10.1007/s00280-021-04308-z. Epub 2021 Jun 7. PMID 34097100